CLINICAL TRIAL: NCT05027698
Title: FEMOSEAL CLOSE - Post-Market Clinical Investigation of the FemoSeal™ VCS: A Prospective, Multi-Center Observational European Study
Brief Title: Post-Market Clinical Investigation of the FemoSeal™ VCS: A Prospective, Multi-Center Observational European Study
Acronym: FEMOSEAL CLOSE
Status: Completed | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T138E4
Record Dates: First submitted 2021-08-13; First posted 2021-08-30 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Vascular Closure; Endovascular Procedure; Hemostasis; Peripheral Vascular Disease
Keywords: peripheral intervention; CFA arteriotomy closure; common femoral artery access site; vascular closure device
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to further demonstrate the safety and effectiveness of the FemoSeal™ VCS in achieving hemostasis following percutaneous endovascular procedures performed via the common femoral artery (CFA) access site. This study is conducted in real-world subjects according to the FemoSeal™ VCS instruction for use (IFU), as part of the study device post-market clinical follow up surveillance plan and prospective clinical evidence collection.

DETAILED DESCRIPTION:
The proposed Post-Market Clinical Follow-up study is a Prospective, Multi-Center, Observational Study, aiming to further demonstrate the safety and effectiveness of the FemoSealTM VCS in achieving hemostasis of common femoral artery (CFA) access site in real-world subjects undergoing percutaneous endovascular procedures. 230 patients will be enrolled at up to 6 European sites. Follow-ups are scheduled at 30 days (±7 days) by hospital visit or telephone call.

The sponsor shall provide training and the necessary guidelines to assist each investigation site on the data collection in the eCRF. Each site is responsible to report the available data requested by the CIP. In order to ensure data quality, validation & consistency, edit checks will be designed during database development. Data Management team and the study monitors will be responsible to review the data and raise queries in the eCRF. Data cleaning will be done in regular intervals specified in Data Monitoring Plan. The final clean standardised datasets will be available prior to database lock for data analysis. An audit trail logging all data entered and edited is available within the EDC system. All source documents are maintained in the hospital files ready for inspection by the Sponsor and regulatory authorities upon request. The Sponsor will inform the investigator of the time period for retaining these records as per applicable regulatory requirements.

The study will be monitored at all stages of its development by study monitors appointed by the sponsor. Study monitors are designated as Sponsor representatives and are assigned to oversee the conduct and progress of the study at each site in accordance with the Monitoring Plan established for this clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years old
2. Subject is willing and able to complete the follow-up requirements
3. Subject has the mental capacity (i.e. does not require the use of a Legally Authorized Representative) to sign the study Informed Consent Form (ICF)
4. Patient undergoing diagnostic or interventional endovascular procedure compatible with the use of FemoSeal™ VCS
5. Puncture site located at the CFA (i.e. between the inferior epigastric artery and the bifurcation of the superficial and profunda femoral arteries)
6. FemoSeal™ VCS deployed as per instruction for use by a trained operator on arteriotomy where sheaths or devices of ≤7F were used, following a femoral artery angiogram

Exclusion Criteria:

1. Any contraindication to the endovascular treatment and/or FemoSeal™ VCS use as per IFU
2. Use of the FemoSeal™ VCS on puncture sites other than CFA
3. Repuncture of the CFA within 90 days at the same access site
4. Enrollment of a patient with the contralateral CFA puncture, when a prior target limb access site has been selected for the study and a FemoSealTM deployment has been performed.

   Additionally, patients will be examined intraoperatively and excluded from the study if any of the following were observed by the treating physician:
5. Lumen diameter of CFA < 5 mm
6. Stenosis and/or significant plaque present in the vicinity of the CFA puncture site
7. Arterial puncture is at, or distal to, the femoral artery bifurcation
8. Anomalous branches or vessel abnormalities present in the vicinity of the CFA puncture site
9. Use of > 7F primary introducer sheaths or devices
10. Multiple femoral punctures
11. Known or suspected posterior femoral wall puncture
12. Any condition that would make use of the closure device inappropriate (as per investigators' discretion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients undergoing diagnostic or interventional endovascular procedures in which FemoSeal™ VCS is used as per it's IFU.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness endpoint: Successful puncture site haemostasis | within 6 hours post procedure
  Cessation of arterial bleeding (excluding oozing) achieved in the CathLab in subjects not requiring any adjunctive intervention at the access site, including (but not limited to) sterile wound dressing and/or manual compression.
Safety endpoint: Freedom from major complications | within 6 hours post procedure
  Freedom from major complications of the access site limb

SECONDARY OUTCOMES:
Freedom from any minor complications at the target limb access site. | within 6 hours post procedure
  Minor complications are defined as:
  * Any puncture site-related haematoma (i.e. a palpable groin swelling measured at the longest diameter)
    * Minor (<5 cm) or
    * Major (≥5 cm)
  * Pseudoaneurysms attributable to the study device
  * Arteriovenous fistulas
  * Minor access site infections (i.e. all infections not defined as major)
Freedom from any major and minor complications at the target limb access site. | within 6 hours to 30 days post-procedure
Time to hemostasis (TTH) | up to 1 day
  Defined as time between the removal of the procedural sheath up to first observed arterial bleeding cessation (excluding oozing at access site) in subjects not requiring adjunctive intervention in the cathlab.
Time to ambulation (TTA) | up to 30 days
  Defined as the time between the procedural sheath removal and the moment when the patient is able to ambulate, i.e. autonomously stand up from the bed and walk without recurrent bleeding.
Length of stay in hospital | up to 30 days
  i. e. the time between the procedural sheath removal and the moment when the patient is discharged from the hospital
Quality of Life assessment | at baseline, discharge , and 30 days
  Quality of Life assessed as per EuroQl five-dimensional (EQ-5D) questionnaire:
  The first part of the questionnaire contain descriptive questions on 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression, each with 5 levels of responses.
  The second part of the questionnaire contains a standard vertical 20-cm visual analog scale that is calibrated from 'the worst health you can imagine' (scored 0) at its base to 'the best health you can imagine' (scored 100) at its apex.
FemoSeal™ VCS usability | up to 1 day
  Accessed by questionnaire, including, but not limited to the following items (usefulness; ease of use; ease of learning; satisfaction and intention to use) completed by operators.

CONTACTS AND LOCATIONS:
Locations (3):
- AZ Sint Blasius, Dendermonde, Belgium
- Hôpital Paris St Joseph, Vascular and endovascular surgical center, Paris, France
- Universitäts-Herzzentrum Freiburg Bad Krozingen, Department of Cardiology and Angiology Department, Bad Krozingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Goueffic Y, Deloose K, Dubosq M, Zeller T. FEMOSEAL CLOSE: multi-centre observational study with FemoSeal vascular closure device following peripheral percutaneous endovascular procedures. CVIR Endovasc. 2025 Feb 22;8(1):15. doi: 10.1186/s42155-025-00522-5. PMID 39985734